CLINICAL TRIAL: NCT00368355
Title: CD-34 Selection for Ex-vivo T-Cell Depletion of Mobilized Peripheral Blood Stem Cells for Recipients of HLA Haploidentical Related Donor Stem Cell Grafts Receiving Intensive Conditioning
Brief Title: T Cell Depletion for Recipients of HLA Haploidentical Related Donor Stem Cell Grafts
Acronym: MOHEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-8701-MOHEL
Record Dates: First submitted 2005-09-21; First posted 2006-08-24 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Acute Lymphoblastic Leukemia; Non Hodgkins Lymphoma; Myelodysplastic Syndrome; Acute Myeloid Leukemia; Chronic Myelogenous Leukemia; Hemophagocytic Lymphohistiocytosis (HLH); Familial Hemophagocytic Lymphohistiocytosis (FLH); Viral-associated Hemophagocytic Syndrome (VAHS); X-linked Lymphoproliferative Disease (XLP)
Keywords: haploidenticalstem cell transplant; acute lymphoblastic leukemia; Non Hodgkins Lymphoma; Myelodysplastic Syndrome; Acute myeloid leukemia; Chronic myelogenous leukemia; Hemophagocytic lymphohistiocytosis (HLH); Familial hemophagocytic lymphohistiocytosis (FLH); Viral-associated hemophagocytic syndrome (VAHS); X-linked lymphoproliferative disease (XLP)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphohistiocytosis, Hemophagocytic; Lymphoproliferative Disorders | interventions — Cytarabine; Cyclophosphamide; Alemtuzumab; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLINIMACS Device (Experimental): Subjects will receive transplant conditioning with Ara-C, Cyclophosphamide, Campath-1H, Total Body Irradiation and will then receive T cell depleted stem cell infusion processed by the CLINIMACS Device
  Interventions: Drug: Ara-C; Drug: Cyclophosphamide; Biological: Campath-1H; Radiation: Total Body Irradiation; Procedure: Stem Cell Infusion
- ISOLEX Device (Experimental): Subjects will receive transplant conditioning with Ara-C, Cyclophosphamide, Campath-1H, Total Body Irradiation and will then receive T cell depleted stem cell infusion processed by the ISOLEX Device
  Interventions: Drug: Ara-C; Drug: Cyclophosphamide; Biological: Campath-1H; Radiation: Total Body Irradiation; Procedure: Stem Cell Infusion

INTERVENTIONS:
Drug: Ara-C — day-8 through day-5
  3 g/m2 q 12 hours
  Other Names: cytarabine
Drug: Cyclophosphamide — day-7 and day-6
  45 mg/kg
  Other Names: Cytoxan
Biological: Campath-1H — day-3 through day-1
  Dosing for children:
  5 - 15kg : 3mg IV in 30ml NS
  15.1 - 30kg : 5mg IV in 50ml NS
  >30 kg : 10mg IV in 100ml NS
  Adults will receive 10mg IV in 100ml NS
  Other Names: Alemtuzumab
Radiation: Total Body Irradiation — day-4 through day-1
  175 cGy x 2 at 24 cGy/min
Procedure: Stem Cell Infusion — Stem cells are infused on day 0

SUMMARY:
Subjects are being asked to participate in this study because treatment of their disease requires them to receive a stem cell transplant. Stem cells or "mother" cells are the source of normal blood cells and lead to recovery of blood counts after bone marrow transplantation (BMT). Unfortunately, there is not a perfectly matched stem cell donor (like a sister or brother) and the subject's disease is considered rapidly progressive and does not permit enough time to identify another donor (like someone from a registry list that is not their relative). We have, however, identified a close relative of the subject's whose stem cells are not a perfect match, but can be used. However, with this type of donor, there is typically an increased risk of developing graft-versus-host disease (GVHD), a high rate of transplant failure, and a longer delay in the recovery of the immune system.

GVHD is a serious and sometimes fatal side effect of stem cell transplant. GVHD occurs when the new donor cells (graft) recognizes that the body tissues of the patient (host) are different from those of the donor. When this happens, cells in the graft may attack the host organs, primarily the skin, liver, and intestines. The number of occurrences and harshness of severe GVHD depends on several factors, including the degree of genetic differences between the donor and recipient, the intensity of the pre-treatment conditioning regimen, the quantity of transplanted cells, and the recipient's age. In recipients of mismatched family member or matched unrelated donor stem cell transplants, there is a greater risk of GVHD so that 70-90% of recipients of unchanged marrow will develop severe GVHD which could include symptoms such as marked diarrhea, liver failure, or even death.

In an effort to lower the occurrences and severity of graft-versus-host disease in patients and to lower the rate of transplant failure, we would like to specially treat the donor's blood cells to remove cells that are most likely to attack the patient's tissues. This will occur in combination with intense conditioning treatment that the patient will receive before the transplant.

DETAILED DESCRIPTION:
To participate in this study, the subject will need to have a central line (a thin plastic catheter or tube that is placed during surgery into one of the large veins in the neck or chest).

Also before treatment can begin, we will test the subject's blood for viruses which can cause problems after the transplant.

Before treatment can begin, stem cells will be collected from the donor that has been selected as the best match for the subject. White blood cells will be collected from the donor. The cells will then be mixed with a special protein called a CD34 antibody that binds to the stem cells which will then be separated out from the white blood cells by a special machine called a CLINIMACs CD34 Reagent System in the laboratory. This is an investigational and experimental device which is not approved by the FDA. Although this device is not approved for use in this country, it has been in use for years and is approved in other countries. The stem cells will be collected and frozen before we start to give chemotherapy.

TREATMENT PLAN

To prepare the subject's body for transplantation, the subject will be given high dose chemotherapy (also called a conditioning treatment) for 8 days prior to the transplant as follows:

The subject will be given a drug called Ara-C in high doses through the central line every 12 hours starting 8 days before transplant (called day - 8) until 5 days before transplant (called day - 5). Starting one day after receiving the first Ara-C dose (day - 7), we will add a drug called cyclophosphamide once a day to the treatment for the next two days. This will be given in high doses (also through the central line). Also on day - 7, we will add a drug called MESNA. MESNA is used to decrease the side effects caused by cyclophosphamide. After the medication treatment is finished (day - 4), radiation treatment will be given to the entire body twice a day for 4 days. The chemotherapy and radiation treatment will last 8 days. If the subject has abnormal cells in the spinal fluid, 6 extra daily doses of radiation treatment may be given to the head. This would be done before any of the drugs are given and before the subject is admitted for transplant.

NOTE: Depending on the subjects health status, the doctor may decide the subject should not receive Ara-C. If this is a possibility, the doctor will discuss this with the subject.

On the second day of radiation (day -3), the subject will receive CAMPATH-1H as a daily 4-hour IV (intravenous, by vein). The subject will receive this infusion once a day for a total of three days. CAMPATH 1H is a special type of protein called an antibody, that works against certain types of blood cells. CAMPATH 1H is important because it stays active in the body for a long time after infusion, which means it may work longer at preventing GVHD symptoms.

The day after the radiation treatment is completed (day 0), the subject will receive the specially selected donor stem cells. Once in the bloodstream, the cells will go to the bone marrow and should begin to grow. If the subject is at risk for developing GVHD or if the subject begins to develop GVHD, the doctor will prescribe medicines to help prevent or treat this side effect. The doctor will describe these medicines at that time.

To learn more about the way the new cells are growing blood will be taken for research purposes at approximately 3 months, 6 months, 9 months, and a year after the transplant. On day 100, the subject will have the same tests/evaluations the subject has been experiencing since the transplant, however, the subject will also have a bone marrow aspirate (we take a sample of bone marrow to evaluate the disease and GVHD status). For patients who do not develop GVHD, they may have an additional bone marrow aspirate on day 180 (about 2 months after the previous one).

After day 365, the subject will be asked to return to the clinic once a year for evaluations. These evaluations will be similar to the ones the subject had on day 100.

ELIGIBILITY:
INCLUSION CRITERIA:

* Lack of suitable conventional donor (i.e. 5/6 or 6/6 related or 5/6 or 6/6 unrelated donor) or presence of a rapidly progressive disease not permitting time to identify an unrelated donor
* Age less than or equal to 55 years of age
* Patients with high risk ALL in CR1 or ALL or high grade (stage III or IV) NHL after first relapse or with primary refractory disease or minimal residual diseases.
* Myelodysplastic syndrome
* Patients with high risk AML in CR1 or after first relapse or with primary refractory disease or minimal residual disease.
* CML
* Hemophagocytic lymphohistiocytosis (HLH), familial hemophagocytic lymphohistiocytosis (FLH), viral-associated hemophagocytic syndrome (VAHS), X-linked lymphoproliferative disease (XLP), Severe chronic active Epstein Barr virus infection (SCAEBV) with predilection for T- or NK-cell malignancy
* Donor cells should be collected and frozen before conditioning starts

EXCLUSION CRITERIA:

* Patients with a life expectancy (< / = 6 weeks) limited by diseases other than leukemia
* Patients with symptomatic cardiac disease, or evidence of significant cardiac disease by echocardiogram (i.e., shortening fraction < 25%)
* Patients with severe renal disease (i.e., creatinine clearance less than 40 cc/1.73 m^2)
* Patients with pre-existing severe restrictive pulmonary disease (FVC less than 40% of predicted)
* Patients with severe hepatic disease (direct bilirubin greater than 3 ug/dl or SGPT (serum glutamic-pyruvic transaminase) greater than 500 ug/dl)
* Patients with severe personality disorder or mental illness
* Patients with a severe infection that on evaluation by the Principal Investigator precludes ablative chemotherapy or successful transplantation
* Patients with documented HIV positivity

'High risk' ALL or AML refers to those acute leukemias identified by the presence of specific biologic features, which predict high likelihood of failure to conventional chemotherapy. As biologic features of high risk disease evolve with improvement of conventional chemotherapy, it is not practical to define this indication with any further specificity. Therefore, high risk AML/ALL will be determined by the primary physician.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2000-04; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Krance, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hosptial, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- CLINIMACS Device: Subjects will receive transplant conditioning with Ara-C, Cyclophosphamide, Campath-1H, Total Body Irradiation and will then receive T cell depleted stem cell infusion processed by the CLINIMACS Device
  Ara-C: day-8 through day-5
  3 g/m2 q 12 hours
  Cyclophosphamide: day-7 and day-6
  45 mg/kg
  Campath-1H: day-3 through day-1
  Dosing for children:
  5 - 15kg : 3mg IV in 30ml NS
  15.1 - 30kg : 5mg IV in 50ml NS
  >30 kg : 10mg IV in 100ml NS
  Adults will receive 10mg IV in 100ml NS
  Total Body Irradiation: day-4 through day-1
  175 cGy x 2 at 24 cGy/min
  Stem Cell Infusion: Stem cells are infused on day 0
- ISOLEX Device: Subjects will receive transplant conditioning with Ara-C, Cyclophosphamide, Campath-1H, Total Body Irradiation and will then receive T cell depleted stem cell infusion processed by the ISOLEX Device
  Ara-C: day-8 through day-5
  3 g/m2 q 12 hours
  Cyclophosphamide: day-7 and day-6
  45 mg/kg
  Campath-1H: day-3 through day-1
  Dosing for children:
  5 - 15kg : 3mg IV in 30ml NS
  15.1 - 30kg : 5mg IV in 50ml NS
  >30 kg : 10mg IV in 100ml NS
  Adults will receive 10mg IV in 100ml NS
  Total Body Irradiation: day-4 through day-1
  175 cGy x 2 at 24 cGy/min
  Stem Cell Infusion: Stem cells are infused on day 0
Period: Overall Study
Arm/Group | CLINIMACS Device | ISOLEX Device
Started | 18 | 28
Completed | 7 | 11
Not Completed | 11 | 17
Not completed — Adverse Event | 1 | 0
Not completed — Death | 2 | 4
Not completed — Relapse | 6 | 10
Not completed — Subsequent transplant | 0 | 3
Not completed — Treatment - hematopoietic cell product | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who had their donor stem cells processed using the ISOLEX or CliniMACS CD34 Reagent System and started preparative regimen were included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | CLINIMACS Device | ISOLEX Device | Total
Number analyzed (Participants) | 18 | 28 | 46
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 7 [5 to 13] | 7 [2.5 to 11] | 7 [3 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 11 | 19 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 5 | 7
  Black or African American | 3 | 8 | 11
  Asian | 1 | 1 | 2
  Hispanic or Latino | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Engraftment Rate After Transplant
Description: Percentage of participants with hematopoietic engraftment post-transplant. Engraftment is defined as the first day absolute neutrophil counts exceeded 0.5 X 10^9/ml.
Time Frame: 28 days
Population: A participant is evaluable for engraftment if the participant underwent transplant and either completed 28 days observation or engrafted. Of the 46 participants at baseline, one in CLINIMACS group did not undergo transplant and one in ISOLEX group died 5 days after transplant.Thus, 2 participants were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CLINIMACS Device | ISOLEX Device
Number analyzed (Participants) | 17 | 27
percentage of participants | 100 [80.5 to 100] | 100 [87.2 to 100]

2. Secondary Outcome: Early Post BMT Toxicities
Description: Number of participants who experience organ failure or severe infections (defined as Grade III/IV by NCI CTC for Adverse Events (CTCAE), version 2.0)
Time Frame: 100 Days
Population: Of the 46 participants at baseline, one participant in CLINIMACS Device group did not undergo haploidentical stem cell transplant and was not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CLINIMACS Device | ISOLEX Device
Number analyzed (Participants) | 17 | 28
Participants | 14 | 14

3. Secondary Outcome: Severe GVHD Rate
Description: Percentage of participants with Grade III/IV acute GVHD. Severe GVHD is defined as Grade III/IV acute GVHD.
Time Frame: 100 Days
Population: A participant is evaluable for acute GVHD if the participant engrafted and either completed 100 days observation after transplant or experienced acute GVHD. Of the 46 participants at baseline, eight participants in CLINIMACS and five in ISOLEX were not evaluable for acute GVHD and were not included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CLINIMACS Device | ISOLEX Device
Number analyzed (Participants) | 10 | 23
percentage of participants | 0 [0 to 30.8] | 4.3 [0.1 to 21.9]

4. Secondary Outcome: Patients With Acute GVHD
Description: Number of participants with acute GVHD graded by the method of Przepiorka et al, which evaluates skin involvement, lower and upper GI, and liver function (bilirubin), each being graded in stages from 0 to 4, where 0 means no acute GVHD, and 4 is the highest stage of acute GVHD
Time Frame: First 100 Days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CLINIMACS Device | ISOLEX Device
Number analyzed (Participants) | 10 | 23
Participants
  Grade 0 | 7 | 16
  Grade I | 3 | 6
  Grade II | 0 | 0
  Grade III | 0 | 0
  Grade IV | 0 | 1

5. Secondary Outcome: Patients With Chronic GVHD
Description: Number of participants with chronic GVHD graded by the method of Przepiorka et al, which evaluates skin, joints, oral, ocular, hepatic, esophagus, GI, respiratory, platelet, and musculoskeletal involvement, in stages from 0 to 3.
Time Frame: Up to 1 Year
Population: Patients surviving more than 100 days were evaluable for chronic GvHD. Of the 46 participants at baseline, eight participants in CLINIMACS and six in ISOLEX were not evaluable for chronic GVHD and were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CLINIMACS Device | ISOLEX Device
Number analyzed (Participants) | 10 | 22
Participants
  No | 10 | 20
  Yes | 0 | 2

6. Other Pre Specified Outcome: Immune Reconstitution
Description: To evaluate the effect of T-cell depletion by positive selection for CD34 on immune reconstitution, which will be determined from total lymphocyte count, from T and B cell numbers and from T cell subset analyses.
Time Frame: 1 Year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Length of Remission in Patients
Description: Median length of remission in patients with high risk leukemia treated with myeloablative chemotherapy, radiotherapy and CD34 selected peripheral blood stem cells from haploidentical related donors using Kaplan-Meier method
Time Frame: 1 Year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time participants started preparative regimen to 100 days post transplant.
Arm/Group | CLINIMACS Device | ISOLEX Device
All-Cause Mortality (participants affected / at risk) | 2/18 | 4/28
Serious Adverse Events (participants affected / at risk) | 14/18 | 15/28
Other Adverse Events (participants affected / at risk) | 13/18 | 23/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLINIMACS Device (N=18) | ISOLEX Device (N=28)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal-Other: Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 0 (0) | 1 (2)
pharyngeal ulcers (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Liver Dysfunction/Failure (clinical) (Hepatobiliary disorders) | 0 (0) | 1 (1)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 0 (0) | 2 (2)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 0 (0) | 1 (1)
Catheter-Related Infection (Infections and infestations) | 2 (3) | 2 (2)
Infection/Febrile Neutropenia-Other: HHV6 viremia (Infections and infestations) | 1 (1) | 0 (0)
Infection(documented clinically or microbiologically)with grade 3 or 4 neutropenia(ANC <1.0 x 10e9/L (Infections and infestations) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 10 (14) | 6 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy - sensory (Nervous system disorders) | 1 (1) | 0 (0)
Adult Respiratory Distress Syndrome(ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary-Other: Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary-Other: Mediastinal hematoma after replacing central line. (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary-Other: Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal/Genitourinary-Other: Hemorrhagic Cystitis (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal/Genitourinary-Other: Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal/Genitourinary-Other: Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLINIMACS Device (N=18) | ISOLEX Device (N=28)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2) | 0 (0)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
GGT (Gamma-Glutamyl transpeptidase) (Investigations) | 0 (0) | 7 (10)
Hepatic enlargement (Hepatobiliary disorders) | 0 (0) | 2 (2)
Portal vein flow (Hepatobiliary disorders) | 1 (1) | 0 (0)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1) | 3 (4)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 3 (7)
Catheter-Related Infection (Infections and infestations) | 2 (2) | 6 (11)
Infection/Febrile Neutropenia -Other: Parainfluenza (Infections and infestations) | 0 (0) | 1 (1)
Infection(documented clinically or microbiologically)with grade 3 or 4 neutropenia(ANC <1.0 x 10e9/L (Infections and infestations) | 9 (10) | 6 (8)
Infection without neutropenia (Infections and infestations) | 2 (2) | 1 (1)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 11 (18)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5) | 3 (4)
Lipase (Investigations) | 0 (0) | 2 (3)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Abdominal Pain or Cramping (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pleural Effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary-Other: Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
BUN (Investigations) | 0 (0) | 1 (1)
Creatinine (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes